CLINICAL TRIAL: NCT01638780
Title: Effect of Resveratrol on Insulin Sensitivity and Metabolic Profile in Type 2 Diabetics
Brief Title: Resveratrol and Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-3-092
Record Dates: First submitted 2012-05-30; First posted 2012-07-12 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Resveratrol; Long-Term Synaptic Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): A placebo will be given for 30 days, twice daily. One pill will be provided with lunch and the other pill will be provided with dinner.
  Interventions: Dietary Supplement: placebo
- resveratrol (Active Comparator): resveratrol will be given for 30 days, twice daily. One pill, which contains 75 mg of resveratrol, will be provided with lunch, and the other pill of 75 mg will be provided with dinner. So in total 150 mg/day of resveratrol will be given.
  Interventions: Dietary Supplement: resveratrol

INTERVENTIONS:
Dietary Supplement: placebo — A placebo will given for 30 days, twice daily. One pill will be provided with lunch, and the other pill will be provided with dinner.
  Arms: placebo
Dietary Supplement: resveratrol — resveratrol will be given for 30 days, twice daily. One pill, which contains 75 mg of resveratrol, will be provided with lunch, and the other pill, also containing 75 mg will be given with dinner. So in total a dose of 150 mg/day will be given.
  Other Names: resVida (99% pure trans-resveratrol) provided by DSM Nutritional Products, Ltd.
  Arms: resveratrol

SUMMARY:
The main objective of the study is to investigate if resveratrol supplementation can improve overall and muscle-specific insulin sensitivity in type 2 diabetic patients.

As a secondary objective the investigators want to investigate whether the improved insulin sensitivity can be attributed to improved muscle mitochondrial oxidative capacity and a reduced intrahepatic and cardiac lipid content.

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* Age: 40-70 years
* Body fat percentage > 25, BMI 27-35 kg/m2
* Diagnosed with type 2 diabetes at least one year before the start of the study
* Well-controlled type 2 diabetics: HBA1C < 8.0%
* Oral glucose lowering medication (metformin only or in combination with sulfonylurea agents)
* Sedentary

  * Not more than 2 hours of sports a week
  * No active job that requires strenuous physical activity
* Stable dietary habits
* Willingness to abstain from resveratrol-containing food products

Exclusion Criteria:

* Unstable body weight (weight gain or loss > 3kg in the last three months)
* Total body fat percentage < 25%
* Hemoglobin < 7.8 mmol/l
* Use of anticoagulants
* Engagement in programmed exercise > 2 hours total per week
* Impaired kidney and/or hepatic function Creatinine 50-100 umol/L Liver enzymes, within 2 times of normal range of laboratory standard (ASAT < 60 U/L, ALAT < 70 U/L, Billi <40 umol/L, gamma-GT < 80 U/L)
* No diabetes related co-morbidities like cardiovascular diseases, diabetic foot, polyneuropathy, retinopathy
* Insulin dependent Diabetic subjects
* Any medical condition except type 2 diabetes mellitus requiring treatment and/or medication use except metformin only or in combination with sulfonylurea agents
* Intake of dietary supplements except multivitamins and minerals
* Current alcohol consumption > 20 grams/day
* Subjects who don't want to be informed about unexpected medical findings during the screening /study, or do not wish that their physician is informed, cannot participate in the study.
* Participation in another biomedical study within 1 month before the first screening visit
* Any contraindication to MRI scanning. These contra-indications include patients with following devices:

  * Central nervous system aneurysm clip
  * Implanted neural stimulator
  * Implanted cardiac pacemaker of defibrillator
  * Cochlear implant
  * Insulin pump
  * Or metal containing corpora aliena in the eye or brains

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2012-05; Primary Completion 2014-09 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
insulin sensitivity (overall, muscle- and liver specific) | 30 days after supplementation

SECONDARY OUTCOMES:
muscle mitochondrial oxidative capacity | 30 days after supplementation
intramyocellular lipid content | 30 days after supplementation
intrahepatic lipid content | 30 days after supplementation
intracardiac lipid content | 30 days after supplementation
heart function | 30 days after supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Silvie Timmers, PhD, Principal Investigator — Human Biology, Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] Timmers S, Konings E, Bilet L, Houtkooper RH, van de Weijer T, Goossens GH, Hoeks J, van der Krieken S, Ryu D, Kersten S, Moonen-Kornips E, Hesselink MKC, Kunz I, Schrauwen-Hinderling VB, Blaak E, Auwerx J, Schrauwen P. Calorie restriction-like effects of 30 days of resveratrol supplementation on energy metabolism and metabolic profile in obese humans. Cell Metab. 2011 Nov 2;14(5):612-22. doi: 10.1016/j.cmet.2011.10.002. PMID 22055504